CLINICAL TRIAL: NCT01136681
Title: Wales Electronic Cohort for Children (WECC)
Brief Title: Wales Electronic Cohort for Children
Acronym: WECC
Status: Completed | Type: Observational
Sponsor: Swansea University (Other)
Collaborators: Cardiff University (Other)
Responsible Party: Principal Investigator, Dr Sarah E. Rodgers, Professor Ronan Lyons, Swansea University
Other Study IDs: TPR08-006
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Macrosomia; Low Birth Weight; Premature Birth; Childhood Obesity; Poverty
Keywords: Anonymised Electronic Cohort; Record Linkage; Routine Data; Environment; Childhood Obesity; Low birth weight; Premature birth
MeSH Terms: conditions — Premature Birth; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators are developing a research platform capable of improving children's health through the generation of knowledge from analysis of routinely collected data from within and outside the health service.

The investigators are using the data that are routinely collected in Wales to answer specific questions about child health and well-being, with the aim of informing policy and practice in Wales, whilst also being internationally relevant.

Routinely collected datasets are publicly funded, and have already been incorporated into the Secure Anonymised Information Linkage databank. The investigators are combining these datasets on children from health and social care to establish an anonymised Wales wide Electronic Cohort for Children (WECC). WECC will serve as the platform for future work in translating information into child population health policy.

There are 35,000 births in Wales per year, and data are available for the previous ten years. Thus, WECC will be sufficiently powered to answer important social, economic and health policy questions. WECC will also act as a demonstration project which would inform the development of e-cohorts to support translational research across the life course and disease spectrum.

DETAILED DESCRIPTION:
Lack of access to the enormous amount of information collected on children's health status and treatment has been a major contributor to both gaps in the translational pathway to improving child health at individual and population levels. The creation of the Wales Electronic Child Cohort is designed to remove this block and support both explanatory and interventional studies. This proposal is considered to be the best way to address this issue as it is built upon previous strategic investments by WORD and thus should achieve its goals in a very cost effective manner.

This type of E-Cohort with 35,000 additional children every year can answer questions where exposures, outcomes and potential confounders are routinely collected or available through individual or ecological linkages. This is a retrospective and prospective cohort, however, both cohort and nested case-control studies can be supported. Developments in geographical information systems (GIS), network analysis and the creation of a system for anonymising households means that is possible to anonymously link environmentally derived data to health data. The huge numbers of individuals involved in WECC means that the study has enormous power to answer important social, economic and health policy questions.

Examples of research questions which can be answered are:

1. What factors determine the future health service need for individuals that are vulnerable at birth, and inform the development of interventions to reduce health inequalities for these groups?
2. What is the influence of the social and physical environment on childhood obesity?
3. What is the impact of health conditions in childhood on educational outcomes for children?
4. Are birth anomalies more common in households in which any member received antibiotics during early pregnancy (marker for infectious cause)?
5. What is the relationship between maternal depression, family composition and childhood injury risk?
6. Can perinatal environmental and biological parameters be used to predict common illness such as asthma in later childhood and adults?
7. To what extent can E-Cohorts replicate findings from traditional cohorts (e.g. Millennium Cohort Study) and replace the need for some non-routine data collection?

In this first instance we will focus on answering the first two questions.

ELIGIBILITY:
Inclusion Criteria:

* Present in routine data and recorded as born or resident in Wales (1998-2008)

Exclusion Criteria:

* Not recorded in routine data as being born of resident in Wales (1998-2008)

Max Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 730,000 children born from 1990-2009, or subsequently resident, in Wales
Sampling Method: Non-Probability Sample
Enrollment: 900000 (Actual)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Birth weight | not applicable due to routine data usage
  Birth weight derived from routine data

CONTACTS AND LOCATIONS:
Overall Officials: Ronan A Lyons, Principal Investigator — Swansea University
Locations (2):
- United Kingdom (2):
  - Health Information Research Unit, Swansea, Swansea
  - Department of Primary Care and Public Health, Cardiff